CLINICAL TRIAL: NCT02368236
Title: Facilitating Risk-Appropriate Colorectal Cancer Testing - Testing the Cancer Risk Intake System (CRIS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 112010-132; R01CA122330 (NIH)
Record Dates: First submitted 2015-01-28; First posted 2015-02-23 (Estimated); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Colorectal Neoplasms; Colonic Neoplasms
Keywords: Early Detection of Cancer; Intervention Studies; Randomized Controlled Trial; Colorectal Neoplasms; Colonic Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intervention Group (Other): Patients randomized to the intervention group will use CRIS. Then intervention group patients and their physicians will receive a tailored printout generated by the CRIS recommending risk-appropriate colorectal testing and ways to overcome perceived barriers to testing. A member of the research team will hand the patient a printout and will deliver the other printout to the physician.
  Interventions: Behavioral: Tailored Printout
- Comparison Group (No Intervention): Patients randomized to the comparison group will use CRIS, but receive a non-tailored standard information about multiple types of cancer screening (e.g., content from an American Cancer Society cancer screening brochure) while physicians receive standard electronic chart prompts indicating the patients were age-eligible but not currently adherent for colorectal cancer screening.
- True No-contact Control Group (No Intervention): A screening baseline for the true no-contact group will be established by conducting a retrospective chart review for patients who did not receive an invitation to participate in this study. The same randomization procedure will be used as the comparison and intervention groups. The purpose is to conduct analysis with the comparison and intervention group to see if individuals who participate in CRIS have a higher screening rate for colorectal cancer compared to the non-contact group.

INTERVENTIONS:
Behavioral: Tailored Printout — The Cancer Risk Intake System (CRIS) is a tablet-based program through which patients answer detailed questions about their colorectal cancer risk prior to an appointment. Tailoring algorithms in CRIS generate printed information for patients and their physicians summarizing their risk factors and matching them with guideline-based screening options.
  Arms: Intervention Group

SUMMARY:
This study will adapt and test a touch-screen computer program to evaluate cancer risk and provide patient-tailored recommendations for appropriate risk-based testing. This individually tailored intervention delivered right at the point of primary care and just prior to the office visit, can be a helpful and non-obstructive adjunct to clinical care.

The primary aim of this project is to test whether a tailored intervention promoting risk-appropriate cancer testing results increases participation compared with a simple non-tailored reminder or no reminder. The trial is designed to determine the extent to which the Cancer Risk Intake System (CRIS) facilitates (1) participation in risk-appropriate colorectal cancer testing, as documented by electronic medical record audit; (2) patient receipt of risk-appropriate colorectal cancer testing recommendations from their physicians, as documented by electronic medical record audit; and (3) changes in patients' intent to participate in risk-appropriate colorectal cancer testing, as documented by patient report.

The Family and Community Medicine and General Internal Medicine clinic databases will be used to identify potentially eligible patients with upcoming scheduled appointments. Because physicians will be the unit of random assignment, patients will be coded before study invitation as potential participants in the intervention or the comparison group. A random sample of eligible intervention and comparison group patients will be selected for contact. Identified patients will be mailed letters from the practices and signed by their physicians requesting their participation. The letters will describe a "study of beliefs and practices about cancer prevention and early detection" and will provide a toll-free number to refuse contact. One week after the mailing, patients who have not called to refuse contact will be called by study staff to explain the study, verify eligibility and, if the patient agrees, to arrange an in-person meeting at the clinic 30 minutes prior to their appointment. These calls will be made by trained research assistants who will follow standard calling protocols. After consent, participants will complete the computerized data collection (CRIS) immediately prior to a scheduled primary-care appointment. Intervention group patients and their physicians will receive a printout recommending risk-appropriate colorectal testing and ways to overcome perceived barriers to testing. A member of the research team will hand the patient his or her printout and will deliver the other printout to the physician. Comparison group patients and physicians will receive non-tailored printouts that are simple reminders about testing.

The investigators will also establish a true no-contact control by conducting a retrospective chart review for randomly selected patients who did not receive an invitation to participate in the study. This no-contact control will establish a baseline screening rate. The investigators will then conduct analysis with the comparison and intervention group to see if individuals who participate in CRIS have a higher screening rate for colorectal cancer compared to the non-contact group. These additional data will help us better assess study Aims 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be considered eligible if they are age 25-75 and have an upcoming appointment and have not had a colonoscopy during the previous 5 years.
* Eligible patients ages 25-49 must also have a family history of colorectal cancer or personal history of inflammatory bowel disease or adenomatous polyps.
* Pregnant women will be included.

Exclusion Criteria:

* Adults younger than age 25 will be excluded because colorectal testing would be inappropriate for the vast majority of patients this young. The benefit of discerning patients in this age group for whom testing would be appropriate would be outweighed by the amount of labor and cost necessary to identify them.
* Patients between ages of 25 and 75 will be excluded if they have had colorectal cancer, a colonoscopy in the last five years, do not give informed consent, do not have access to a telephone, or have severely impaired hearing or speech.
* In addition, patients between ages 25 and 49 will be excluded unless they have a close relative diagnosed with Colon or Rectal Cancer before the age of [pts age + 11] or they've had a colon polyp or inflammatory bowel disease.
* Patients who do not speak or read English will not be eligible for participation in the main study. In years 3 and 4, patients whose main language is Spanish will be included for participation in cognitive interviews and a pilot test to ensure the S-CRIS is culturally appropriate, conceptually equivalent, and usable for the diverse Spanish-speaking primary-care population.
* Patients who are cognitively impaired will be excluded from all parts of the study.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1012 (Actual)
Dates: Start 2008-12; Primary Completion 2012-02 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Participation in risk-appropriate colorectal cancer testing (i.e., participation in any CRIS-recommended test based on patients' risk factors). | 12 month post baseline
  Mixed-effects logistic regression model. Group assignment = main independent variable. Physician = random cluster effect.
  Binary outcome values:
  * Participation in any risk-appropriate CRIS-recommended test.
  * Either no testing or participation in a non-recommended test (e.g., stool-based test for an individual whose risk profile indicated need for colonoscopy).
  For patients assigned to the:
  * Intervention group (i.e., tailored printout).
  * Comparison group (i.e., non-tailored printout).

SECONDARY OUTCOMES:
Participation in any type of colorectal cancer testing. | 12 month post baseline
  Mixed-effects logistic regression model. Group assignment = main independent variable. Physician = random cluster effect.
  Binary outcome values:
  * Participation in any testing.
  * No participation in testing within 12 months.
  For patients assigned to the:
  * Intervention group (i.e., tailored printout).
  * Comparison group (i.e., non-tailored printout).
Testing difference in receipt of any type of colorectal cancer testing. | 12 month post baseline
  Mixed-effects logistic regression model. Group assignment = main independent variable. Physician = random cluster effect. Age and gender = covariates.
  Difference between patients assigned to:
  * Use CRIS (i.e., intervention group = tailored printout and comparison group = non-tailored printout).
  * True no-contact control group.

CONTACTS AND LOCATIONS:
Overall Officials: Celette S Skinner, PhD, Principal Investigator — University of Texas Southwestern Medical Center

IPD SHARING:
Plan to Share IPD: No